CLINICAL TRIAL: NCT03812562
Title: Pilot Study of Nivolumab in Combination With Therasphere (Yttrium-90) for Treatment of Hepatocellular Carcinoma (HCC) With Intent for Resection
Brief Title: Nivolumab and Yttrium-90 in Treating Patients With Liver Cancer Undergoing Surgical Resection
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Northwestern University (Other)
Collaborators: Bristol-Myers Squibb (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 18I03; NU 18I03 (Other: Northwestern University); NCI-2018-03602 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA060553 (NIH)
Record Dates: First submitted 2019-01-16; First posted 2019-01-23 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (yttrium Y 90 glass microspheres, nivolumab) (Experimental): Patients receive standard of care yttrium Y 90 glass microspheres IV. Within 1-2 weeks of completing of yttrium-90 treatment, patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 4 doses in the absence of disease progression or unacceptable toxicity. If imaging shows adequate FLR and at least stable disease, patients will undergo resection within 2 weeks after the last dose of nivolumab. Patients who do not complete resection due to feasibility and have progressed or have evidence of high-risk explant may continue to receive nivolumab IV every 2 weeks for up to 1 year.
  Interventions: Biological: Nivolumab; Radiation: Yttrium Y 90 Glass Microspheres

INTERVENTIONS:
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Yttrium Y 90 Glass Microspheres — Given IV
  Other Names: TheraSphere

SUMMARY:
This early phase I trial studies how well nivolumab and yttrium-90 work in treating patients with liver cancer who are undergoing surgical resection. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radioactive drugs, such as yttrium-90, may carry radiation directly to tumor cells and not harm normal cells. Giving nivolumab and yttrium-90 may work better in treating patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the hepatocellular carcinoma (HCC) recurrence rate post-resection in patients intended to undergo resection post yttrium Y 90 glass microspheres (yttrium-90 [Y-90]) + nivolumab.

SECONDARY OBJECTIVES:

I. To investigate the safety and feasibility of radioembolization and nivolumab in patients with HCC with intent for resection.

II. To assess the pattern of recurrence post-resection (time frame and location of recurrence).

III. To evaluate efficacy in patients with HCC treated with Y90 + nivolumab using overall survival.

IV. To evaluate the drop-out rate and incremental changes in future liver remnant (FLR).

EXPLORATORY OBJECTIVES:

I. To assess immune-related biomarkers from original tumor biopsy if available. II. To identify differences in immunological profiles among patients who go undergo resection versus those who do not undergo resection due to progression or failure to grow FLR to sufficient level. III. In patients with hepatitis C virus (HCV), will explore changes in immunological profile associated with direct acting anti-viral agents.

OUTLINE:

Patients receive standard of care yttrium Y 90 glass microspheres intravenously (IV). Within 1-2 weeks of completing of yttrium-90 treatment, patients receive nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks for up to 4 doses in the absence of disease progression or unacceptable toxicity. If imaging shows adequate FLR and at least stable disease, patients will undergo resection within 2 weeks after the last dose of nivolumab. Patients who do not complete resection due to feasibility and have progressed or have evidence of high-risk explant may continue to receive nivolumab IV every 2 weeks for up to 1 year.

After completion of study treatment, patients are followed up at 30 days and then periodically for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of hepatocellular carcinoma (HCC) confirmed by American Association for Study of Liver Diseases (AASLD) guidelines with a Childs-Pugh score of A or B (but, =< Childs score B8)
* Patients must be eligible for resection based on preserved hepatic function and lack of clinically significant portal hypertension (HTN)

  * NOTE: Patients with branch or lobar portal vein thrombosis (PVT) who are otherwise a candidate for resection will be included
* Patients must have a pre-established need for Y90 therapy prior to resection for FLR growth and/or retraction of tumor away from major vessel to improve margins
* Patients must have measurable disease according to the standard Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Patients with chronic hepatitis B are eligible as long as they have evidence of ongoing viral replication (detectable hepatitis B surface antigen [HBsAg], hepatitis B e-antigen [HBeAg], or hepatitis B virus [HBV] deoxyribonucleic acid [DNA]). They must have HBV DNA viral load < 100 IU/mL at screening. In addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy. If not on antiviral therapy at screening, then the subject must initiate treatment per regional standard of care guidelines at the time of consent. Both HBeAg positive and negative patients will be included
* Patients positive for hepatitis C are permitted at physician discretion
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Adequate organ and bone marrow functions:
* Leukocytes >= 2,000/mcL
* Absolute neutrophil count >= 1,500/uL
* Hemoglobin >= 9 g/dL; transfusion is permitted for eligibility, but should be >= 7 days from registration
* Platelets >= 50,000/mcL
* Total bilirubin =< 2.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Serum creatinine of =< 2.0 x ULN (upper limit of normal) or creatinine clearance >= 30 mL/minute (using Cockcroft/Gault formula below):

  * Female creatinine clearance (CrCl) = (140 - age in years) x weight in kg x 0.85/ 72 x serum creatinine in mg/dL
  * Male CrCl = (140 - age in years) x weight in kg x 1.00/ 72 x serum creatinine in mg/dL
* Females of childbearing potential (FOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) =< 7 days prior to registration

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

    * Has not undergone a hysterectomy or bilateral oophorectomy
    * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
  * NOTE: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* FOCBP and men who are sexually active with FOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and the designated post-treatment period
* Ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy =< 28 days prior to registration are not eligible
* Patients who have had prior immunotherapy including interleukin-2 and immune checkpoint antagonist and/or agonists are not eligible
* Patients who have not recovered to their baseline, =< grade 1, or tolerable grade 2 (as documented by the treating physician) from adverse events due to agents administered >= 28 days earlier are not eligible
* Patients who have received any other investigational agents =< 28 days prior to registration are not eligible
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab or Y90 are not eligible
* Patients who have had prior treatment with an anti-PD1, anti-PD-L1, antiPD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways are not eligible
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including chronic prolonged systemic corticosteroids (defined as corticosteroid use of duration one month or greater), should be excluded. These include but are not limited to patients with a history of:

  * Immune related neurologic disease
  * Multiple sclerosis
  * Autoimmune (demyelinating) neuropathy
  * Pure red cell aplasia
  * Guillain-Barre syndrome
  * Myasthenia gravis
  * Systemic autoimmune disease such as systemic lupus erythematosus (SLE)
  * Connective tissue diseases
  * Scleroderma
  * Inflammatory bowel disease (IBD)
  * Crohn?s
  * Ulcerative colitis
  * Patients with a history of toxic epidermal necrolysis (TEN)
  * Stevens-Johnson syndrome
  * Anti-phospholipid syndrome

    * NOTE: Subjects with vitiligo, alopecia, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Patients with any condition requiring systemic treatment with corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications =< 14 days prior to registration are not eligible

  * NOTE: Inhaled steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. A brief (less than 3 weeks) course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by a contact allergen) is permitted
* Patients who have received live vaccine =< 28 days from registration are not eligible

  * NOTE: Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist) are live attenuated vaccines, and are not allowed at any time during the study
* Patients with uncontrolled intercurrent illness including, but not limited to any of the following, are not eligible:

  * Hypertension that is not controlled on medication
  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient?s safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* Patients with new brain metastases are not eligible unless they have had treatment of lesions and are neurologically stable off steroids prior to registration
* Patients with another primary malignancy within 2 years of registration are not eligible with the following exceptions: adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix, or any localized cancers that are deemed to be cured from investigator?s point of view
* Patients with known history of human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are not eligible
* Prisoners or participants who are involuntarily incarcerated are not eligible

  * NOTE: under certain specific circumstances a person who has been imprisoned may be included as a participant. Strict conditions apply and Bristol-Myers Squibb approval is required)
* Participants must not be compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Recurrence rate | Up to 3 years post-treatment
  This primary dichotomous endpoint will be summarized at each time point using a table of frequencies and counts.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days post-treatment
  Incidence of adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Will be tabulated and reviewed.
Overall survival (OS) | Up to 5 years post-treatment
  OS distributions will be estimated using the Kaplan Meier method, with estimates for the 25th percentile, median and 75th percentile for each time-to-event outcome. In addition, specific Kaplan-Meier estimates for survival at 1-year will be calculated, with Greenwood?s formula for variance used to calculate a 95% confidence interval (CI).
Overall increase in future liver remnant (FLR) | Up to 3 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kulik, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States